CLINICAL TRIAL: NCT05170893
Title: Efficacy and Safety of Coenzyme Q10 in Pediatric Hemodialysis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Salma AbdelRahman, Principal Investigator, Misr International University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: ACUC-FP-ASU RHDIRB2020110301
Record Dates: First submitted 2021-12-11; First posted 2021-12-28 (Actual); Last update posted 2023-07-19 (Actual); Status verified 2023-07

CONDITIONS: Hemodialysis
MeSH Terms: interventions — coenzyme Q10; Ubiquinone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Oral Coenzyme Q10 capsules daily for 12 weeks.
  Interventions: Dietary Supplement: Coenzyme Q10
- Control group (Placebo Comparator): Oral capsules similar to the intervention daily for 12 weeks.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Coenzyme Q10 — Oral capsules
  Other Names: ubiquinone, ubidecarenone, ubiquitous quinone
  Arms: Intervention group
Other: Placebo — Oral capsules
  Arms: Control group

SUMMARY:
All chronic kidney disease patients, whether on regular hemodialysis or not, are at high risk of cardiovascular diseases. This is mainly due to increased oxidative stress, reduced antioxidants and generalized inflammation. Coenzyme Q10 is a vitamin-like antioxidant synthesized in almost all body cells, and it is also available in many dietary sources. It was observed that chronic kidney disease patients have low plasma levels of Coenzyme Q10. Clinical benefits of Coenzyme Q10 supplementation have been documented for various cardiovascular and neurodegenerative disorders. The investigators believe that Coenzyme Q10 supplementation may have potential benefits in pediatric patients receiving hemodialysis; mainly due to its antioxidant activity and anti-inflammatory effects.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients with ages between 2 to 18 years old.
* Undergoing regular hemodialysis for at least 6 months.

Exclusion Criteria:

* Patients who weigh less than 10 kg.

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 36 (Actual)
Dates: Start 2022-01-17 (Actual); Primary Completion 2022-07-14 (Actual); Study Completion 2022-07-26 (Actual)

PRIMARY OUTCOMES:
Change in Malondialdehyde (MDA) | 12 weeks
  marker of oxidative stress

CONTACTS AND LOCATIONS:
Locations (1):
- El-Demerdash Children's Hospital, Cairo, Egypt